CLINICAL TRIAL: NCT07075991
Title: The Uptake and Excretion of a Single Oral Dose of 1 µm [14C]-Labelled Polystyrene Microplastic Particles in Healthy Volunteers Using a Micro Dose Approach
Brief Title: Uptake and Excretion of a Single Dose of Oral 14C-labelled Polystyrene Microplastics in Healthy Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); TNO (Other)
Responsible Party: Principal Investigator, Marlou Dirks, Assistant Professor, Wageningen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL88025.028.25
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Kinetics
Keywords: Microplastics; Uptake; Excretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): [14C]-labelled PS-MP ingestion
  Interventions: Drug: 1 μm [14C]-labelled Polystyrene Microplastic

INTERVENTIONS:
Drug: 1 μm [14C]-labelled Polystyrene Microplastic — A single test day during which participants will orally ingest a single micro dose of 100 μg 1 µm [14C]-labelled PS-MP. Prior to and following ingestion of the labelled PS-MP, biological samples (i.e. blood, urine, faeces) will be collected at regular intervals, throughout the 5-day study period. Participants will spend the first 24h in the clinical laboratory, after which they are allowed to spend the remainder of the 5-day study period at home but with daily visits to the laboratory for blood sampling and home collection of urine and faeces.

SUMMARY:
The goal of this clinical trial is to understand how a small, labeled dose of microplastics moves through the human body (i.e., how it is absorbed, distributed, and excreted) in healthy adult volunteers aged 18-65 years (3 males, 3 females). The main questions it aims to answer are:

* How much of the ingested microplastic is absorbed into the bloodstream?
* How is the microplastic distributed and eliminated from the body through urine and feces?

Participants will:

* Take a single oral micro dose of 100 µg of 1 μm [14C]-labelled polystyrene microplastics (PS-MP).
* Spend 24 hours in a clinical research facility for close monitoring and initial sample collection.
* Provide blood, urine, and stool samples over a 5-day period (with daily short lab visits after the first day).

This study does not include a comparison group.

DETAILED DESCRIPTION:
Human exposure to micro- and nanoplastics (MNPs) is increasingly recognized, yet their internal behavior in the body-absorption, distribution, and elimination-is still not well understood. No human data currently exist to support toxicokinetic modeling, which is essential for translating laboratory (in vitro) data into risk assessments. This study addresses this gap by quantifying the biokinetics of a single oral microdose of 1 μm [14C]-labelled polystyrene microplastics in healthy volunteers. By using Accelerator Mass Spectrometry (AMS), extremely low concentrations of radiolabeled particles can be accurately measured in biological matrices (blood, urine, and feces). This will provide critical benchmark data to validate in vitro-to-in vivo extrapolations and improve human health risk assessments for microplastics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females using contraception during and for 3 months after the study.
* Aged from 18-65 years at the time of signing informed consent
* 18.5 < BMI < 25 kg·m-2
* Must be willing and able to communicate and participate in the whole study
* Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)

Exclusion Criteria:

* Diabetes (Type 1, Type 2, or genetic form of diabetes)
* Any diagnosed cardiovascular (heart) disease or high blood pressure (≥140 mmHg systolic and/or ≥90 mmHg diastolic)
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastro-intestinal disease, immunodeficiency, endocrine, neurological or psychiatric disorders
* Known severe kidney problems
* Subjects who have regular gastrointestinal complaints including abdominal pain, stomach upsets and borborygmi, known or suspected irritable bowel syndrome, or functional constipation
* Recent or chronic history of diarrhoea
* Known anaemia
* Known impaired liver function
* A personal or family history of thrombosis (clots), epilepsy, seizures, or schizophrenia.
* Chronic use of any prescribed or over the counter pharmaceuticals (excluding oral contraceptives and contraceptive devices)
* History of any drug or alcohol abuse in the past two years
* A confirmed positive alcohol breath test at screening or admission
* Any known food allergies or intolerances to the 14 major food allergens (celery, cereals containing gluten, crustaceans, eggs, fish, lupin, milk, molluscs, mustard, tree nuts, peanuts, sesame seeds, soybeans, sulphur dioxide and sulphites) or history of a malabsorption syndrome including coeliac disease
* Currently taking part in other scientific research
* Having received a product with 14C in the past 12 months
* Pregnant or breastfeeding
* Subjects who have taken antibiotics within the 60 days prior to the adaptation period.
* Unable to give consent
* Employed or undertaking a thesis or internship at the department of Human and Animal Physiology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Biokinetic profile (absorption, distribution, excretion) of [14C]-labelled PS-MP | 5 days post-administration
  Quantitative assessment of 14C content in blood, urine, and feces using Accelerator Mass Spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Department of Human and Animal Physiology, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request to the Principal Investigator